CLINICAL TRIAL: NCT02629029
Title: Multi-Modality Imaging for Head & Neck Cancer Free Flap Design and Assessment
Brief Title: Multi-Modality Imaging for Head & Neck Cancer Free Flap Design Assessment
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We are closing this study due to the focus on other research projects and there is no time or personnel tofurther pursue the completion of this project
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-8151
Record Dates: First submitted 2015-06-01; First posted 2015-12-11 (Estimated); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Contrast Media; Computed Tomography Angiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Surgical - therapeutic free flap (Other): patients will be enrolled under informed consent based upon their medical diagnosis, planned surgical procedures, and suitability for the procedure. During the study, patients will be imaged using two systems: (i) pre-operative CTA with IV contrast; (ii) intra-operative fluorescence endoscopy with ICG.
  Interventions: Procedure: Pre-op CTA with IV contrast; Device: Computed tomography angiography (CTA)

INTERVENTIONS:
Procedure: Pre-op CTA with IV contrast — Preoperative mapping of perforators by computed tomography angiography (CTA) could prove valuable in head and neck free flap transfer and shorten the operation time significantly. This modality could provide useful information for H&N cancer reconstruction in difficult cases, especially in patients with large or through-and-through defects that might need multiple perforators in flap design. In addition, near-infrared (NIR) fluorescence imaging using indocyanine green (ICG) angiography can provide robust, intraoperative, objective data to optimize the free flap skin paddle design while potentially minimizing patient morbidity.
  Other Names: Intra-operative fluorescence endoscopy with ICG
Device: Computed tomography angiography (CTA)

SUMMARY:
Surgical reconstruction of anatomical structures after head and neck cancer resection has made enormous strides in the past 20 years with advancing flap techniques and the usage of perforating vessels, but accurate and consistent identification of these perforators has remained a challenge due to the varying anatomy of vasculature in the donor region. Computed tomography angiography (CTA) has been used increasingly in preoperative free flap perforator mapping for breast reconstruction but has been limited in head and neck applications. In addition, indocyanine green (ICG) assisted NIR fluorescence angiography has been developed for intra-operative flap assessment. In this study, the investigators propose to assess a previously undocumented, multi-modal imaging technique with preoperative dual energy CTA to design and intraoperative ICG assisted NIR angiography to assess free flap in head and neck reconstruction.

DETAILED DESCRIPTION:
CTA and NIR-assisted ICG angiography will be used in the mapping of the free flaps. CTA provides surgeons with preoperative information on the vascular anatomy and facilitates surgical planning for flap harvesting. The advantages of CTA are that it is noninvasive, rapid, and easy to read by the surgeon. Moreover, it provides information to help the surgeon decide which site to explore in the operation and reduces the rate of injuring or missing an optimal perforator.

This technique can help reduce the size of the incision needed for perforator exploration, which helps reduce the patient's postoperative discomfort. The operation time can be reduced by choosing suitable perforators in the preoperative stage, which can also help reduce the cost of hospitalization. NIR-assisted angiography gives live localization of the flap's dominant perforator perfusion zones while quantifying the relative tissue perfusion for immediate skin paddle design.

ELIGIBILITY:
Inclusion Criteria:

* The study will include patients planned for free anterolateral thigh/fibula or scapula flap for Head&Neck cancer reconstruction.
* The patients should have a complete and detailed medical record.
* Subjects must be at least 18 years of age.
* Subjects must sign and be given a copy of the written Informed Consent Form.

Exclusion Criteria:

* Patients who are not able to consent by themselves or grasp the implication of the study.
* Subjects participating in any other clinical trial during the time of this clinical investigation and that may have an impact on this evaluation.
* Pregnant or potentially pregnant woman
* Lactation.
* Iodine, shellfish, cough mixture, betadine or ICG allergy
* The exclusion criteria for the IV contrast detailed in appendix 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-05-30 (Actual); Primary Completion 2020-11-27 (Actual); Study Completion 2020-11-27 (Actual)

PRIMARY OUTCOMES:
Flap perforators for harvesting | During surgical procedure
  to assess the performance of dual-energy computed tomography and near-infrared fluorescence angiography in evaluating the perforators of a head and neck free flap preoperative and intraoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Irish, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada